CLINICAL TRIAL: NCT04336475
Title: The Effect of a Combined Home-based Orofacial Exercise Program on Oral Aperture of Patients With Systemic Sclerosis: a Single-blind Prospective Randomized Controlled Trial
Brief Title: The Effect of a Home-based Orofacial Exercise Program on Oral Aperture of Systemic Sclerosis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Nihan Cüzdan, Principal Investigator, Cukurova University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Cukurova University Nihan C.
Record Dates: First submitted 2020-04-03; First posted 2020-04-07 (Actual); Results first posted 2020-04-29 (Actual); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: Microstomia; Systemic Sclerosis
Keywords: exercise; microstomia; oral aperture; rehabilitation; systemic sclerosis
MeSH Terms: conditions — Microstomia; Scleroderma, Systemic; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): exercise regimen and oral hygiene care advices
  Interventions: Other: orofacial exercise program
- Group 2 (Active Comparator): oral hygiene care advices
  Interventions: Other: orofacial exercise program

INTERVENTIONS:
Other: orofacial exercise program — combined stretching&strengthening exercise regimen

SUMMARY:
Systemic sclerosis is a systemic disease which may involve multiple organ systems and cause functional disabilities. Microstomia is one of the most common complications of the disease which may result in difficulties performing oral self-care, complication in professional dental care and even malnutrition in the advanced cases. Since the disease is rare and the studies are limited, there is still not an agreed upon orofacial exercise program to improve the oral aperture of the patients. Therefore, we aimed to investigate the effect of a newly diseased home-based exercise program for improving microstomia in those patient population.

DETAILED DESCRIPTION:
The study was designed as a single-blind, prospective, randomized controlled study with a 2-month follow-up period, carried out in rheumatology outpatient clinic, between March 2017 - January 2019. Systemic sclerosis patients with an oral aperture of <40mm were included in the study. Patients were randomly divided into two groups. Randomization was done as the sealed envelope method. After the informed consent was taken, the opaque envelope that the patient have chosen was opened and patients were offered the allocated treatment regimen. Group 1 was given exercise regimen and oral hygiene care advices for the first one month; followed by no exercise but oral hygiene care advices for the next four weeks. Group 2, as the control group, received oral hygiene care advices for the first one month, followed by the exercise regimen twice a day along with oral hygiene care advices for the next four weeks. Oral care advices were given to every participant by a dentist involved in the study at their first visit. With this protocol, we aimed (a) to investigate whether there is a benefit of the exercise program on microstomia; (b) to observe the carryover effect of exercise therapy on microstomia after discontinuing the treatment over a period of time; (c) to estimate the intervention strategy by comparing the same medical approach with different sequences. The exercise program was demonstrated to patients by a clinician at the first visit and given to all patients printed as a manual to be done every day for one month duration of the exercise program. Additionally, a diary was given to patients to mark when they have completed the exercise and to note in the case of pain on daily basis. The exercise regimen was developed on the basis of previous studies and clinical knowledge.

ELIGIBILITY:
Inclusion Criteria:

* systemic sclerosis patients with an interincisal distance of <40 mm

Exclusion Criteria:

* patients with missing teeth
* dysfunction of temporo-mandibular joints
* oral malignancy
* recent dental procedures
* multiple active digital ulcers
* diagnosed psychiatric conditions

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nihan Cuzdan, MD, Principal Investigator — MD
Locations (1):
- Cukurova University, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD may be shared with other researches.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: up to 6 months
Access Criteria: researchers who are willing to access to individual participant data will be reviewed and approved by the principal investigator.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited based on randomization in outpatient rheumatology clinic. First patient was enrolled on March 2017 and the last participant was enrolled in October 2018.
Pre-assignment Details: 156 patients were evaluated and 74 met inclusion criteria. 14 patients refused to participate. 60 patients were randomized.
Groups:
- Exercise + Oral Hygiene First, Then Oral Hygiene Only: Each exercise should be performed two times per day for 5 repetitions, holding each 10 seconds for one month duration in addition to oral hygiene care. After the first month, patients continue only with daily oral hygiene care. Exercise regimen includes: 1.The subject stretches the lips with fingers. 2. The subject inflates the cheeks. 3.The subject keeps maximal mouth opening. 4. The subject bites a wood stick with right & left molars. 5.The subject pushes the chin to left and right sides.
- Oral Hygiene Only First, Then Exercise + Oral Hygiene: patients only perform daily oral hygiene care advices for the first month. Patients start performing exercise program in addition to oral hygiene care advices in the second month. Each exercise should be performed two times per day for 5 repetitions, holding each 10 seconds. 1.The subject stretches the lips with fingers. 2. The subject inflates the cheeks. 3.The subject keeps maximal mouth opening. 4. The subject bites a wood stick with right & left molars. 5.The subject pushes the chin to left and right sides.
Period: Overall Study
Arm/Group | Exercise + Oral Hygiene First, Then Oral Hygiene Only | Oral Hygiene Only First, Then Exercise + Oral Hygiene
Started | 30 | 30
Completed | 28 | 28
Not Completed | 2 | 2
Not completed — pain | 1 | 0
Not completed — upper respiratory infection | 1 | 0
Not completed — Lost to Follow-up | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exercise + Oral Hygiene First, Then Oral Hygiene Only | Oral Hygiene Only First, Then Exercise + Oral Hygiene | Total
Number analyzed (Participants) | 28 | 28 | 56
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 22 | 24 | 46
  >=65 years | 6 | 4 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.82 (9.63) | 50.0 (11.4) | 52 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 26 | 53
  Male | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 28 | 28 | 56
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Turkey | 28 | 28 | 56
oral aperture [Mean (Standard Deviation); unit: milimeters] — interincisal distance between the maxillary and mandibular central incisors in the midline. Patients were asked to open their mouth as wide as they could in the natural head position. The linear distance from the incisal edge of the upper central incisor to the incisal edge of the lower central incisor was recorded using a dental bow compass and measured using a millimeter ruler. Each subject was measured three times every two minutes and the highest value of these three measurements was recorded as millimeters.
  milimeters | 31.17 (4.90) | 33.05 (5.53) | 32.11 (5.26)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Oral Aperture Measurement
Description: the interincisal distance between the maxillary and mandibular central incisors in the midline
Time Frame: 2 months
Measure: Mean (Standard Deviation); unit: milimeters
Groups:
- Exercise + Oral Hygiene First, Then Oral Hygiene Only: 1. st month > exercise + oral hygiene
  2. nd month> oral hygiene only
- Oral Hygiene Only First, Then Exercise + Oral Hygiene: 1. st month> Oral Hygiene Only
  2. nd month > exercise + oral hygiene
Arm/Group | Exercise + Oral Hygiene First, Then Oral Hygiene Only | Oral Hygiene Only First, Then Exercise + Oral Hygiene
Number analyzed (Participants) | 28 | 28
milimeters
  1 st month | 32.98 (5.01) | 32.92 (6.13)
  2 nd month | 33.40 (5.33) | 34.37 (6.47)
Statistical Analysis 1: Comparison: Exercise + Oral Hygiene First, Then Oral Hygiene Only vs Oral Hygiene Only First, Then Exercise + Oral Hygiene; Test type: Superiority; p = 0.564, ANOVA — The threshold for statistical significance was p=0.05. p value stands for the comparison of final oral aperture measurements between two groups. (after 2 months' period); Repeated Measures ANOVA

ADVERSE EVENTS:
Time Frame: 2 months
Description: since this is not a drug study mortality and serious adverse events are not expected.
Groups:
- Exercise + Oral Hygiene: Each exercise should be performed two times per day for 5 repetitions, holding each 10 seconds for one month duration in addition to oral hygiene care.
- Oral Hygiene Only: Patients only perform daily oral hygiene care advices
Arm/Group | Exercise + Oral Hygiene | Oral Hygiene Only
All-Cause Mortality (participants affected / at risk) | 0/56 | 0/56
Serious Adverse Events (participants affected / at risk) | 0/56 | 0/56
Other Adverse Events (participants affected / at risk) | 1/56 | 0/56
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exercise + Oral Hygiene (N=56) | Oral Hygiene Only (N=56)
pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-06-10): https://cdn.clinicaltrials.gov/large-docs/75/NCT04336475/Prot_SAP_000.pdf
  • Informed Consent Form (2016-06-10): https://cdn.clinicaltrials.gov/large-docs/75/NCT04336475/ICF_001.pdf